CLINICAL TRIAL: NCT01434706
Title: NAT: The Early Test Program: Implementation of NAT Screening to Identify Acute and Early HIV Infection at San Diego Public HIV Counseling and Testing Sites
Brief Title: Implementation of Nucleic Acid Amplification Testing Screening to Identify Acute and Early HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Davey Smith, MD, MAS, Professor of Medicinie, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-1414
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Acute HIV Infection
Keywords: HIV; acute infection; primary infection; seroconverters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nucleic Acid Amplification Testing (Other): Nucleic Acid Amplification Testing
  Interventions: Other: Nucleic Acid Amplification Testing

INTERVENTIONS:
Other: Nucleic Acid Amplification Testing — The Gen-Probe Transcription-Mediated Amplification (TMA) technology exponentially amplifies captured HIV-1 and HCV RNA in blood samples. The Gen-Probe system is available in two commercially available FDA approved products; 1) the Procleix assay is a multiplex system that is used to screen the blood supply for HIV and HCV. This assay will allow the simultaneous detection of all known HIV-1 subtypes with sensitivities designed to reduce the window period of false negative results from standard HIV antibody testing (EIA), while maintaining the ability to discriminate positive from negative specimens, even at very low copy numbers (Giachetti, Linnen et al., 2002).

SUMMARY:
The investigators propose to study the impact of nucleic acid amplification testing (NAT) screening for acute Human Immunodeficiency Virus (HIV) and Hepatitis C (HCV) infections and Less-Sensitive Enzyme linked Immunoassay (LS-EIA) or 'detuned' testing Vironostika, Trinity Biotech BED, or Ortho-Clinical Diagnostic Vistros ECi for early HIV infection in conjunction with routine rapid HIV testing at HIV counseling and testing sites and venues in the San Diego county. The overarching goal of this study is to develop and implement a system to identify, notify and engage into care those individuals with recent HIV infection in order to better define the HIV and Hepatitis C Virus (HCV) epidemics in the San Diego county and to evaluate and characterize HIV transmission dynamics within the San Diego population.

ELIGIBILITY:
Inclusion Criteria:

* Persons presenting for HIV testing to Public Health Department HIV testing site.
* Men and women >13 years of age.
* Those who are 13 or older and younger than 18 should be an emancipated minor or have consent given by their legal representative.
* Participants 18 and over must be able to provide written consent.
* Participants should be available for follow up for a period of at least 2 weeks after enrollment

Exclusion Criteria:

* Refusal to participate.
* Unable to provide informed consent.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22607 (Actual)
Dates: Start 2010-09-16 (Actual); Primary Completion 2015-04-07 (Actual); Study Completion 2015-04-07 (Actual)

PRIMARY OUTCOMES:
Nucleic Acid Amplification Testing | 10 minutes
  Positive detection of presence of HIV

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Christie's Place, San Diego, California
  - San Diego LGBT Community Center, San Diego, California
  - UC San Diego Antiviral Research Center, San Diego, California
  - UCSD Lead the Way Storefront, San Diego, California
  - Family Health Centers of San Diego, San Diego, California

REFERENCES:
- See also: The Early Test — https://theearlytest.ucsd.edu/